CLINICAL TRIAL: NCT01007890
Title: Prediction of Response to Neoadjuvant Chemotherapy in Women With Operable Breast Cancer
Acronym: PT-304
Status: Terminated | Type: Observational
Sponsor: Precision Therapeutics (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: PT-304
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Breast Cancer
Keywords: ChemoFX; Operable; Breast; Cancer; Measurable; Disease
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Core needle biopsy specimens will be collected and stored in RNAlater® until the time of RNA extraction, using standard procedures. Isolated total RNA will be assayed for gene expression using methods such as TaqMan® RT-PCR technology or Affymetrix or Agilent gene array platforms.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: ChemoFX Assay — Test of an algorithm to predict pathologic response in patients treated with neoadjuvant chemotherapy for breast cancer.

SUMMARY:
The objective of this study is to develop a biomarker to predict pathological complete response in women treated with neoadjuvant chemotherapy for breast cancer. Such a biomarker would assist physicians in selecting the most effective chemotherapy for the individual patient.

DETAILED DESCRIPTION:
The objective of this study is to develop a biomarker to predict pathological complete response in women treated with neoadjuvant chemotherapy for breast cancer. Such a biomarker would assist physicians in selecting the most effective chemotherapy for the individual patient. The anticipated biomarker will take into account clinical factors (such as tumor stage, tumor size, and age), phenotypic characteristics of the tumor (determined by pathological immunohistochemistry and ex vivo ChemoResponse assay), and genotypic characteristics of the tumor and patient (determined by genomic profiling via gene expression analysis of tumor RNA). It is expected that collective consideration of all of these factors will be more predictive of patient response to therapy than any of them alone.

Approximately 224 evaluable subjects will be recruited from approximately 30 US sites. Women with measurable operable invasive breast cancer diagnosed by core needle biopsy will be eligible for this study. Additional tumor specimens will be obtained prior to the start of chemotherapy via core needle biopsies to be used for the ex vivo ChemoResponse Assay and tumor genomic analysis (gene expression), respectively.

All subjects will receive neoadjuvant chemotherapy with one of two standard of care regimens that must consist of the following agents: doxorubicin (A), cyclophosphamide (C), and a taxane (T) such as docetaxel, paclitaxel, or Abraxane (nanoparticle albumin-bound paclitaxel [nab-paclitaxel]); or, docetaxel (T) and cyclophosphamide (C). These must be administered per NCCN guidelines by the treating physician.

Upon completion of chemotherapy treatment, women will undergo lumpectomy, modified radical mastectomy or other surgical procedure determined appropriate by the investigator and at that time will be evaluated for pathological response. At the time of lumpectomy, modified radical mastectomy, or other surgical procedure, additional tumor excess will be sent to Precision Therapeutics, Inc. (Precision) for exploratory analysis if there is no pathologic complete response (pCR), if there are sufficient tumor cells to send, and if the patient agrees to have her excess tumor cells sent to Precision for this purpose.

During the patient's course of participation on the study, the treating physician will remain blinded to the results of the ChemoResponse Assay and genomic analysis. If it is determined there is no pCR at the time of lumpectomy, modified radical mastectomy or other surgical procedure, Precision will make available a subsequent report to the physician containing additional information about chemotherapy drugs other than ACT that could benefit the further treatment decisions for the patient.

ELIGIBILITY:
Inclusion Criteria

Female subjects who satisfy the following conditions will be considered for enrollment into the study:

1. The subject must consent to be in the research study and must have signed an approved consent form conforming to institutional guidelines prior to study entry.
2. The diagnosis of breast cancer can be made by FNA or biopsy (other than incisional or excisional). The tumor specimen must demonstrate a diagnosis of invasive adenocarcinoma.
3. The primary breast cancer must be operable and measurable "greater than or equal to" 2.0 cm by use of physical exam and/or ultrasound, MRI, CT scan, or mammogram.
4. T1c, T2, T3, or T4 patients clinically staged as M0 (non-inflammatory) are eligible.
5. Patients with a prior diagnosis and treatment for DCIS are eligible.
6. Patients with multi-focal breast cancer are eligible.
7. The tumor must be confined to either the breast or to the breast and ipsilateral axilla.
8. The subject must be 18 years or older.
9. The interval between initial cytologic or histologic diagnosis of breast cancer and registration must be no more than 10 weeks.
10. ECOG Performance Status of 0 or 1 (see Appendix A) is required.
11. The subject must receive standard of care chemotherapy regimens consisting of either doxorubicin (A), cyclophosphamide (C), and a taxane (T) such as docetaxel, paclitaxel, or nab-paclitaxel administered in any sequence and combination the treating physician determines or docetaxel (T) plus cyclophosphamide (C).

Exclusion Criteria

Male subjects are not eligible for this study as the incidence of breast cancer in male subjects is significantly lower than female subjects. Those subjects who are strongly HER2-positive will be excluded as they will require treatment by biological agents for which the ChemoResponse Assay has not yet been validated. Subjects with evidence of distant metastatic disease are excluded as these subjects would not be good candidates for neoadjuvant therapy. Women who have had an excisional or incisional biopsy prior to entry would not have sufficient tumor sample to test or to be measured by physical exam for the study. Women who have nonmalignant comorbid conditions and diseases that would preclude them from being treated with doxorubicin (A), cyclophosphamide (C), and a taxane (T), and from completing the study are also excluded. Women with psychiatric or addictive disorders are excluded to protect those vulnerable subjects who may not be able to adequately give informed consent.

Women with one or more of the following conditions will be ineligible for this study:

1. Tumor determined to be strongly HER2-positive by immunohistochemistry (3+) or by fluorescent in situ hybridization (positive for gene amplification)
2. Definitive clinical or radiologic evidence of distant metastatic disease.
3. Excisional or incisional biopsy for this primary breast tumor.
4. Inflammatory breast cancer.
5. Synchronous contra-lateral breast cancer.
6. Multi-centric breast cancer.
7. Participation in the NSABP B-40 study.
8. Prior therapy for invasive breast cancer, including irradiation, chemo-, immuno-, and/or hormonal therapy.

   a. Note: the only exception is hormonal therapy, which may have been given anytime after diagnosis and before study entry as long as the hormonal therapy is discontinued at or before registration. After surgery, hormonal therapy may be re-started, at the discretion of the treating physician.
9. Current therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulator (SERM), either for osteoporosis or breast cancer prevention, or sex hormonal therapy such as birth control pills, ovarian hormonal replacement therapy, etc. These patients are eligible IF these medications are discontinued prior to registration.
10. Surgical axillary staging procedure prior to study entry.

    a. Note: exceptions include FNA of an axillary node and pre-neoadjuvant sentinel lymph node biopsy for patients with clinically negative axillary nodes.
11. Nonmalignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude the woman from being treated with doxorubicin (A), cyclophosphamide (C), and a taxane (T), and from completing the study.
12. Psychiatric or addictive disorders that would preclude obtaining informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women 18 years or older with Palpable Operable Breast Cancer Measurable Disease
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Primary clinical endpoint pCR will be a dichotomous outcome variable with two levels: complete response and no complete response. | 24 months

SECONDARY OUTCOMES:
Secondary clinical endpoint cOR will be an ordinal outcome variable with complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) four levels. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Lis, RN, MSN, Study Director — Precision Therapeutics
Locations (28):
- United States (28):
  - Breastlink Medical Group, Inc, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Advanced Medical Specialties, Miami, Florida
  - Advanced Breast Care, Marietta, Georgia
  - Missouri Cancer Associates, Columbia, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Breast Care, Las Vegas, Nevada
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Beth Israel Medical Center, New York, New York
  - OU Medical Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Breast Care Specialists, P.C., Allentown, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Breast Clinic of Memphis, Germantown, Tennessee
  - Advantage Clinical Research, Nashville, Tennessee
  - Tennessee Breast Specialists, Nashville, Tennessee
  - Texas Oncology - Bedford, Bedford, Texas
  - Dallas Surgical Group, Dallas, Texas
  - Leading Edge Research, PA, Dallas, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Southlake Oncology, Southlake, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin